CLINICAL TRIAL: NCT00449241
Title: Acupuncture Treatment in Adults Undergoing Diagnostic Upper Gastrintestinal Endoscopy: A Double-Blind Placebo Controlled Randomized Trial
Brief Title: Acupuncture Treatment in Adults Undergoing Diagnostic OGD : A Double-Blind Placebo Controlled Randomized Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRE-2006.227-T
Record Dates: First submitted 2007-03-19; First posted 2007-03-20 (Estimated); Last update posted 2007-03-20 (Estimated); Status verified 2007-03

CONDITIONS: Anxiety
Keywords: Acupuncture, Endoscopy
MeSH Terms: conditions — Anxiety Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Acupuncture

SUMMARY:
To find out how the application of acupuncture needles to the proposed acupuncture points: Heart 7 (HT 7) and Pericardium 6 (PC 6) for reducing anxiety during Esophago-gastro-duodenoscopy (EGD)

DETAILED DESCRIPTION:
Acupuncture is being used as one part of Chinese medicine for more than 2,500 years in treating diseases. Recent functional magnetic resonance imaging demonstrated that acupuncture can suppress the "pain" area in the brain so as to reduce the pain that felt by human subjects. Western medicine proposed the acupuncture mechanisms as to "provoke the release of endogenous substances" from central nervous system so in reducing pain. Many studies had been done using acupuncture in reducing pain for post-operation period, however, most of them were not very systematic and even some of them are leak of control group. Furthermore, to our knowledge, the use of acupuncture for reducing anxiety during EGD has not been previously investigated.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 undergoing elective unsedatant diagnostic EGD
* belonging to American Society of Anesthesia (ASA) classes 1 to 2

Exclusion Criteria:

* History of gastrectomy, esophagectomy, Whipple's operation and other gastrointestinal operations
* ASA class 3 to 4
* Pregnancy
* Allergy to acupuncture needles
* Request sedation
* Previous experiences of EGD

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210
Dates: Start 2006-11; Study Completion 2007-07 (Estimated)

PRIMARY OUTCOMES:
Anxiety elicited during EGD

SECONDARY OUTCOMES:
Overall tolerance, overall satisfaction, patient's willingness to repeat procedure and recovery time

CONTACTS AND LOCATIONS:
Overall Officials: Wing Wa Leung, Master, Principal Investigator — Department of Surgery, CUHK
Locations (1):
- Combined Endoscopy Centre, Alices Ho Miu Ling Netherole Hospital, Hong Kong, China